CLINICAL TRIAL: NCT02698579
Title: Long-term Follow-up of Subjects With Cerebral Adrenoleukodystrophy Who Were Treated With Lenti-D Drug Product
Brief Title: Long-term Follow-up of Participants With Cerebral Adrenoleukodystrophy Who Were Treated With Lenti-D Drug Product
Status: Active, not recruiting | Type: Observational
Sponsor: Genetix Biotherapeutics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LTF-304; 2024-513904-33-00 (EU CTIS Number); 2015-002805-13 (EudraCT Number)
Record Dates: First submitted 2016-02-17; First posted 2016-03-03 (Estimated); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Adrenoleukodystrophy (CALD); Adrenoleukodystrophy (ALD); X-Linked Adrenoleukodystrophy (X-ALD)
Keywords: Adrenoleukodystrophy; X-linked Adrenoleukodystrophy; Hematopoietic Stem Cells
MeSH Terms: conditions — Adrenoleukodystrophy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Long-term followup: Participants who have received Lenti-D Drug Product in a parent clinical study (bluebird bio-sponsored clinical studies ALD-102 and ALD-104) and who meet the eligibility criteria for the Study LTF-304 will be followed in this long-term followup study for 13 years (for a total of 15 years of follow-up after drug product infusion in the parent studies).
  Interventions: Genetic: No interventional drug product utilized in this follow-up study

INTERVENTIONS:
Genetic: No interventional drug product utilized in this follow-up study — Participants received a single IV infusion of Lenti-D Drug Product (also known as elivaldogene autotemcel or eli-cel) in either parent Study ALD-102 or ALD-104.
  The objectives of this long-term follow-up study are to assess long-term safety and efficacy following completion of participation in parent studies. Vector copy number (VCN) measurement, safety evaluations, disease-specific assessments, and assessments to monitor for long-term complications of autologous transplant are conducted in this study.

SUMMARY:
This is a multi-center, long-term safety and efficacy follow-up study for participants with cerebral adrenoleukodystrophy (CALD) who have received Lenti-D Drug Product (eli-cel) in a parent clinical study (Study ALD-102 or Study ALD-104).

After completing a parent clinical study (approximately 2 years), eligible participants will be followed for an additional 13 years for a total of 15 years post-drug product infusion. No investigational drug product will be administered in this study.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent for this study by the participant or participant's parent(s)/ legal guardian(s) and written informed assent by participant, if applicable
* Have received eli-cel in a parent clinical study

Exclusion Criteria:

* There are no exclusion criteria for this study

Max Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Participants with cerebral adrenoleukodystrophy (CALD) who have received Lenti-D Drug Product in a parent clinical study will be expected to participate in this long-term follow-up study.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2016-01-22 (Actual); Primary Completion 2038-08 (Estimated); Study Completion 2038-08 (Estimated)

PRIMARY OUTCOMES:
Major functional disability (MFD)-free survival | 15 years post-drug-product infusion
  The MFDs are loss of communication, cortical blindness, tube feeding, total incontinence, wheelchair dependence, complete loss of voluntary movement.
Number of participants with malignancies | 15 years post-drug-product infusion
Number of participants who experience graft versus host disease (GVHD) | 15 years post-drug-product infusion
Number of participants with immune-related adverse events (AEs) | 15 years post-drug-product infusion
Number of participants with new or worsening hematologic disorders | 15 years post-drug-product infusion
Number of participants with new or worsening neurologic disorders | 15 years post-drug-product infusion

SECONDARY OUTCOMES:
Number of participants who undergo subsequent stem cell transplantation | 15 years post-drug-product infusion
Change from baseline in neurological function score (NFS) | 15 years post-drug-product infusion
  The NFS is a 25-point score used to evaluate the severity of gross neurologic dysfunction in CALD by scoring 15 symptoms (functional domains) across 6 categories. Listed here are the 15 symptoms followed by their maximal score out of 25 points: a) Hearing / auditory processing problems-1, b) Aphasia / apraxia-1, c) Loss of communication-3, d) Vision impairment /field cut-1, e) Cortical blindness-2, f) Swallowing / other central nervous system (CNS) dysfunctions-2, g) Tube feeding-2, h) Running difficulties / hyperreflexia-1, i) Walking difficulties / spasticity / spastic gait (no assistance)-1, j) Spastic gait (needs assistance)-2, k) Wheelchair dependence-2, l) Complete loss of voluntary movement-3, m) Episodes of incontinence -1, n) Total incontinence-2, o) Nonfebrile seizures-1. A score of "0" denotes absence of clinical signs of cerebral disease. Maximal signs within a domain score the total of all grades within that domain.
Number of participants without gadolinium enhancement (GdE) status on magnetic resonance imaging (MRI) | 15 years post-drug-product infusion
  Contrast enhancement (gadolinium enhancement; GdE+) on brain MRI represents a clinically important radiographic biomarker of active neuroinflammatory disease and poor prognosis (in untreated patients). As such, assessment of the number of participants who remained negative for gadolinium enhancement (GdE-) was conducted for this outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Vinod K Prasad, MD, FRCP, Study Director — bluebird bio, Inc.
Locations (13):
- United States (4):
  - Mattel Children's Hospital-UCLA, Los Angeles, California
  - Lucile Packard Children's Hospital - Stanford, Palo Alto, California
  - Boston Children's Hospital/Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
- Instituto Neurogenia, Caba, Argentina
- Women's and Children's Hospital, North Adelaide, Australia
- Hospital das Clínicas da Universidade de São Paulo, São Paulo, Brazil
- Hôpital Bicêtre, Le Kremlin-Bicêtre, Cedex, France
- Universitätsklinikum Leipzig AöR, Leipzig, Germany
- Ospedale Pediatrico Bambino Gesù, Rome, Italy
- Prinses Maxima Center, Utrecht, Netherlands
- United Kingdom (2):
  - Royal Free London Hospital, London, England
  - Great Ormond Street Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
bluebird bio is committed to transparency. Appropriately de-identified patient-level datasets and supporting documents may be shared following attainment of applicable marketing approvals associated with this study and consistent with criteria established by bluebird bio and/or industry best practices to maintain the privacy of study participants. For enquiries, please contact us at datasharing@bluebirdbio.com.

REFERENCES:
- [Derived] Eichler F, Duncan CN, Musolino PL, Lund TC, Gupta AO, De Oliveira S, Thrasher AJ, Aubourg P, Kuhl JS, Loes DJ, Amartino H, Smith N, Folloni Fernandes J, Sevin C, Sankar R, Hussain SA, Gissen P, Dalle JH, Platzbecker U, Downey GF, McNeil E, Demopoulos L, Dietz AC, Thakar HL, Orchard PJ, Williams DA. Lentiviral Gene Therapy for Cerebral Adrenoleukodystrophy. N Engl J Med. 2024 Oct 10;391(14):1302-1312. doi: 10.1056/NEJMoa2400442. PMID 39383459
- [Derived] Duncan CN, Bledsoe JR, Grzywacz B, Beckman A, Bonner M, Eichler FS, Kuhl JS, Harris MH, Slauson S, Colvin RA, Prasad VK, Downey GF, Pierciey FJ, Kinney MA, Foos M, Lodaya A, Floro N, Parsons G, Dietz AC, Gupta AO, Orchard PJ, Thakar HL, Williams DA. Hematologic Cancer after Gene Therapy for Cerebral Adrenoleukodystrophy. N Engl J Med. 2024 Oct 10;391(14):1287-1301. doi: 10.1056/NEJMoa2405541. PMID 39383458
- See also: Parent Study ALD-102 protocol registrations and summary result disclosure — https://clinicaltrials.gov/study/NCT01896102
- See also: Parent Study ALD-104 protocol registrations and summary result disclosure — https://clinicaltrials.gov/study/NCT03852498